CLINICAL TRIAL: NCT05748626
Title: Do Anti-Snoring Appliances Reduce the Amount of Airway Manipulation in Patients Undergoing Anesthetic Sedation? A Prospective Randomized Controlled Trial
Brief Title: Anti-Snoring Appliances and Airway Manipulation in Patients Undergoing Anesthetic Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mahesh Vaidyanathan, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00218263
Record Dates: First submitted 2022-11-14; First posted 2023-03-01 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Airway Obstruction; Snoring; Sedation Complication
Keywords: Airway obstruction; Snoring; Monitored Anesthesia Care; Intravenous sedation
MeSH Terms: conditions — Airway Obstruction; Snoring

STUDY DESIGN:
Intervention Model Description: Randomized controlled interventional trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group #1: Anti-snoring appliance (Experimental): Group #1: Anti-snoring appliance (Zyppah) that will be utilized during their procedure.
  Interventions: Device: Anti-snoring device
- Group #2: Control group, that will not utilize anti-snoring appliance (Active Comparator): Group #2: Control group, that will not utilize (Zyppah) anti-snoring appliance during their procedure.
  Interventions: Procedure: No anti -snoring device during their procedure.

INTERVENTIONS:
Device: Anti-snoring device — For group 1, the study team will aid the subject in molding and preparing the device in the pre-operative area. They will wear the device throughout the entirety of the case.
  Arms: Group #1: Anti-snoring appliance
Procedure: No anti -snoring device during their procedure. — For group 2 there will be no anti snoring device used during the case.
  Other Names: No intervention
  Arms: Group #2: Control group, that will not utilize anti-snoring appliance

SUMMARY:
Would patients using an anti-snoring appliance intraoperatively require less airway manipulation, interventions, and rescue maneuvers during anesthetic sedation cases compared to those who do not? The investigators will use anti-snoring appliance devices (specifically the FDA approved Zyppah) to attempt to relieve tissue obstructions that cause snoring during sleep. The application of the devices to the body is less invasive than other common intraoperative rescue airway devices (e.g. nasal trumpets and oral airways) which are not designed to be patient specific.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18-89 years old)
* Undergoing procedures below the umbilicus requiring anesthetic sedation without an invasive airway
* a STOP-BANG (survey) score of 2 or greater.

Exclusion Criteria:

* Patients who are unable to consent
* Non-English speaking
* Those requiring general anesthesia.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Vaidyanathan, MD,MBA, Principal Investigator — Northwestern Univesity
Locations (1):
- Northwestern Memorial Hospital and Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lacquiere DA, Hodzovic I, Woollard A, Varvinskiy A, Chishti K, Hughes R. DAS 2015 guidelines for management of CICO. Br J Anaesth. 2016 Oct;117(4):532-533. doi: 10.1093/bja/aew285. No abstract available. PMID 28077547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 7 | 4 | 11
Age, Continuous [Median (Full Range); unit: Years] | 66.5 [38 to 84] | 63.2 [50 to 80] | 64.8 [38 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Chicago, Illinois, United States
  participants
    United States | 12 | 13 | 25
Height (Inches) [Mean (Standard Deviation); unit: Inches] | 66.0 (4.2) | 68.1 (4.0) | 67 (4.5)
Weight (Kilograms) [Mean (Standard Deviation); unit: Kilograms] | 89.3 (19.6) | 90 (18.3) | 89.6 (19.1)
Body Mass Index [Mean (Standard Deviation); unit: (kg) / height (m)^2] | 31.8 (6.9) | 30.0 (5.2) | 30.88 (5.88)
American Society of Anesthesiology Status [Count of Participants; unit: Participants] — American Society of Anesthesiology (ASA PS Score) system used to classify a patient's physical health prior to surgery. The score, ranges from I to VI (with an added "E" for emergencies), indicates the severity of a patient's systemic disease.
  ASA I: Healthy patient. ASA II: Mild systemic disease. ASA III: Severe systemic disease. ASA IV: Severe systemic disease that is a constant threat to life. ASA V: Moribund patient who is not expected to survive without the operation. ASA VI: Brain Dead (donor) E: Add E if the patient requires emergency surgery.
  Participants
    ASA 2 Status | 9 | 5 | 14
    ASA 3 Status | 3 | 8 | 11
Documented Mallampati Score [Count of Participants; unit: Participants] — Mallampati score is used in anesthesiology to assess the visibility of structures in the mouth (soft palate, uvula, faucial pillars) and predict the difficulty of intubation. A higher score is associated with a higher likelihood of difficult intubation.
  Class I: Soft palate, uvula, and faucial pillars are completely visible. Class II: Soft palate and uvula are visible, but the faucial pillars are partially or completely masked.
  Class III: Soft palate is visible, but the uvula is masked, and only the base of the uvula may be visible.
  Class IV: Only the hard palate is visible.
  Participants
    Mallampati Score Class 1 | 2 | 5 | 7
    Mallampati Score Class 2 | 5 | 4 | 9
    Mallampati Score Class 3 | 4 | 3 | 7
    Mallampati Score Class 4 | 1 | 1 | 2
Documented Obstructive Sleep Apnea [Count of Participants; unit: Participants] — Documented sleep apnea recorded in the electronic medical record.
  Participants | 0 | 0 | 0
STOP Bang Score [Mean (Standard Deviation); unit: Score on Scale (0 low risk -8 high risk)] — STOP Bang tool is used to assess the risk of obstructive sleep apnea (OSA). based on a questionnaire with eight yes/no questions, and the total score (ranging from 0 to 8) indicates the likelihood of having moderate to severe OSA. A higher score suggests a greater risk of OSA.
  Score on Scale (0 low risk -8 high risk) | 3.3 (.8) | 3.0 (.8) | 3.14 (.8)

OUTCOME MEASURES:

1. Primary Outcome: Combined Total Number of Airway Interventions During an Anesthetic Sedation Case
Description: Combined total number of airway interventions during an anesthetic sedation case - including head tilt/rotation, mandible thrust, chin lift, shoulder lift, neck extension or flexion, tongue pull.
Time Frame: Through study completion, an average of 1 day
Measure: Number; unit: Airway Interventions
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Airway Interventions | 7 | 5

2. Secondary Outcome: Maximum End-tidal CO2
Description: Maximum end-tidal CO2 using measures the partial pressure or maximal concentration of carbon dioxide (CO2) at the end of an exhaled breath, which is expressed as a percentage of CO2 or mmHg. The normal values are 5% to 6% CO2, which is equivalent to 35-45 mmHg.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 41 (9.4) | 44.4 (5.5)

3. Secondary Outcome: Number of Instances SpO2 Value < 92%
Description: Number of instances the SpO2 drops below 92% during the procedure
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Episodes | .6 (.9) | .1 (.3)

4. Secondary Outcome: Minimum End-title CO2 in mmHg
Description: Minimum end-tidal CO2 (capnography) using measures the partial pressure or maximal concentration of carbon dioxide (CO2) at the end of an exhaled breath, which is expressed as a percentage of CO2 or mmHg. The normal values are 5% to 6% CO2, which is equivalent to 35-45 mmHg.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 7 (7.4) | 6.7 (5.0)

5. Secondary Outcome: Percent Time During the Case the SpO2 is Below 92%
Description: Percent time during the case the SpO2 is below 92% using pulse oximetry.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Percent of Time
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Percent of Time | .7 (1.2) | .1 (.3)

6. Secondary Outcome: Maximum SpO2 Value During the Case
Description: Maximum SpO2 value during the case using pulse oximetry (percent saturated)
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Percent | 99.9 (.3) | 99.5 (1.7)

7. Secondary Outcome: Minimum SpO2 Value During the Case
Description: Minimum SpO2 value during the case using pulse oximetry (percent saturation)
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Percent | 91.3 (5.9) | 94.8 (3.0)

8. Secondary Outcome: Heart Rate Maximum
Description: Maximum heart rate during case using standard operating room cardiac monitor
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Heart Rate (Beats Per Minute)
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Heart Rate (Beats Per Minute) | 80.8 (14.3) | 82.5 (15)

9. Secondary Outcome: Heart Rate Minimum
Description: Minimum heart rate during case using standard operating room cardiac monitor
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Heart Rate (Beats Per Minute)
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Heart Rate (Beats Per Minute) | 53.4 (6.5) | 58.5 (11.1)

10. Secondary Outcome: Maximum Systolic Blood Pressure
Description: Maximum systolic blood pressure (mmHg) using standard operating room blood pressure cuff and monitor.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 140 (16.9) | 152.2 (21.7)

11. Secondary Outcome: Minimum Systolic Blood Pressure
Description: Minimum systolic blood pressure (mmHg) using standard operating room blood pressure cuff and monitor.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 88.9 (9.1) | 88.1 (13.7)

12. Secondary Outcome: Maximum Diastolic Blood Pressure
Description: Maximum diastolic blood pressure (mmHG) using standard operating room blood pressure cuff and monitor.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 75.3 (14.3) | 77.1 (8.7)

13. Secondary Outcome: Minimum Diastolic Blood Pressure
Description: Minimum diastolic blood pressure (mmHG) using standard operating room blood pressure cuff and monitor.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 51.2 (5.1) | 53.2 (14.7)

14. Secondary Outcome: Minimum Mean Blood Pressure
Description: Mean minimum diastolic blood pressure (mmHG) using standard operating room blood pressure cuff and monitor.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 65.1 (6.4) | 64.6 (9.2)

15. Secondary Outcome: Maximum Mean Blood Pressure
Description: Maximum mean blood pressure (mmHG) using standard operating room blood pressure cuff and monitor.
Time Frame: Through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
mmHG | 98.4 (12.5) | 104.5 (15.6)

16. Secondary Outcome: Reintubation in the Post Anesthesia Care Unit
Description: Number of participants requiring reintubation with an endotracheal tube post surgery in the Post Anesthesia Care Unit
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

17. Secondary Outcome: Surgical Length of Time
Description: Surgical length of time in hours.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
Number analyzed (Participants) | 12 | 13
Hours | 2.5 (.5) | 2.6 (.4)

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Group #1: Anti-snoring Appliance | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 1/12 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group #1: Anti-snoring Appliance (N=12) | Group #2: Control Group, That Will Not Utilize Anti-snoring Appliance (N=13)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cough in the Post Anesthesia Care Unit
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Bronchospasm in the Post Anesthesia Care Unit
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) — Regurgitation event in Post Anesthesia Care Unit
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Aspiration of gastric contents into the airway in the PACU
Case converted to general anesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Surgical case changed to general anesthesia during the procedure due to respiratory deficiency.
Rapid Response Team Alerted (Cardiac disorders) | 0 (0) | 0 (0) — Rapid Response Team alerted for cardiac and or respiratory failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT05748626/Prot_SAP_001.pdf